CLINICAL TRIAL: NCT06675409
Title: Comparing Expert Guided Training and Self -Directed Learning with Virtual Patients in Emergency Management Training : a Randomized Controlled Trial
Brief Title: Expert Guided Training Versus Self Learning with Virtual Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Dilek Kitapçıoğlu, Assist Prof., Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Acibadem U
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-08

CONDITIONS: Educational Problems; Virtual Patient; Emergencies
Keywords: virtual patient; emergency patient management; self directed learning
MeSH Terms: conditions — Emergencies | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Expert Guided Group (Active Comparator): The expert-guided group will participate in virtual patient sessions consisting of 12 patient scenarios under the guidance of an expert. These patient scenarios are selected clinical cases designed to enhance critical decision-making skills in emergency patient management. Throughout the training, students will receive verbal feedback from experts on their performance
  Interventions: Other: Education
- Self Learning Group (Experimental): The self-learning group will also participate in training with the same 12 patient scenarios as the other group, but instead of expert guidance, the students in this group will engage with the virtual patient scenarios independently and manage the process without instructor guidance. In this group, feedback on students' performance will be provided in written form by the computer-based virtual patient simulator.
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — The effectiveness of two different training methods with virtual patients for improving the critical decision-making skills of paramedic students will be compared between two groups: one receiving expert-guided training and the other following a self-directed approach

SUMMARY:
Virtual patients have increasingly been used in the training of healthcare professionals to enhance critical decision-making skills in emergency patient management education. The aim of this study is to investigate the contribution of the virtual patient simulation used in the education of paramedic students by comparing the effectiveness of self-directed learning with expert-guided learning. Additionally, it is believed that the study will be beneficial for educators responsible for program design who are interested in integrating the case-based learning method with virtual patients into their curriculum.

DETAILED DESCRIPTION:
Virtual patient-based simulation training is increasingly being used in healthcare and medical education to enhance problem-solving and critical decision-making skills. There are two common approaches in these trainings: instructor-led learning and self-directed learning. In instructor-led virtual patient-based simulation training programs, an experienced subject matter expert guides students through virtual patient simulation activities. The instructor provides feedback, support, and encourages discussion and collaboration among students during the training. This approach is beneficial for students who benefit from structured activities and social support in a group learning environment. However, it can be time-consuming, costly, and may not be suitable for every student.

In self-directed learning, the responsibility for learning lies entirely with the student. Students are given access to virtual patient simulations and are encouraged to work through the cases independently. This approach may be more suitable for students who are self-motivated, enjoy autonomy, and have the discipline to work independently. It also offers a cost-effective and flexible option. However, in this approach, the feedback and support needed for skill development are limited to the feedback reports generated by the computer-based virtual patient software program.

In the literature, studies on the use of virtual patient applications in paramedic students' emergency patient management training are limited. This study aims to contribute to educators who use or plan to use virtual patient simulation by comparing instructor-led virtual patient-based simulation training with self-directed virtual patient-based simulation training to determine which approach is more effective in enhancing students' critical decision-making skills.

ELIGIBILITY:
Inclusion Criteria:

Volunteer 4th-semester paramedic students from the Department of Vocational Health Sciences at the University

Exclusion Criteria:

Previous experience with the same clinical scenarios

Ages: 19 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Virtual patient exam scores of the participants | 1 week
  All the participants will attend to the virtual patient exam and the scores will be compared between groups

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem Mehmet Ali Aydinlar University CASE Simulation Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No